CLINICAL TRIAL: NCT02914158
Title: Adjuvant Ovarian Suppression Plus Aromatase Inhibitor or Tamoxifen for Hormone Receptor-Positive Breast Cancer in Women Younger Than 35: A Multicenter Randomized Clinical Trial
Brief Title: Adjuvant Ovarian Suppression Plus Aromatase Inhibitor or Tamoxifen in Young Women
Acronym: ASPAIT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Ying Lin, Vice Director of Department of Breast Surgery, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20160818GD
Record Dates: First submitted 2016-09-18; First posted 2016-09-26 (Estimated); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; ovarian function suppression (OFS); aromatase inhibitors（AIs）; tamoxifen（TAM）
MeSH Terms: conditions — Breast Neoplasms | interventions — Goserelin; Tamoxifen; Aromatase Inhibitors; Leuprolide

ARMS (2):
- Ovarian Suppression and aromatase inhibitors (Experimental): Ovarian Suppression：Goserelin 3.6 mg or Leuprolide 3.75 mg administered intravenously every 28 days, for 5 years.
  AI: no restriction of specific drugs, oral by standard dose of post-menopause breast cancer, for 5 years.
  Interventions: Drug: Goserelin; Drug: Aromatase Inhibitors; Drug: Leuprolide
- Ovarian Suppression and tamoxifen (Active Comparator): Ovarian Suppression：Goserelin 3.6 mg or Leuprolide 3.75 mg administered intravenously every 28 days, for 5 years.
  Tamoxifen: 20mg oral for every day, for 5 years.
  Interventions: Drug: Goserelin; Drug: Tamoxifen; Drug: Leuprolide

INTERVENTIONS:
Drug: Goserelin
Drug: Tamoxifen
  Arms: Ovarian Suppression and tamoxifen
Drug: Aromatase Inhibitors
  Arms: Ovarian Suppression and aromatase inhibitors
Drug: Leuprolide
  Other Names: leuprolide acetate

SUMMARY:
The objective of this study is to compare the curative effects in patients under the age of 35 with hormone receptor positive breast cancer and high recurrent risk factors including large tumor or metastatic lymph nodes randomized to ovarian function suppression (OFS) plus aromatase inhibitors or OFS plus tamoxifen as adjuvant endocrine therapy, and explore the differences of curative effects between different subtypes to provide direct evidence for treatments of young breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent;
2. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2;
3. Patients pathologically diagnosed with hormone receptor positive invasive breast cancer: immunohistochemistry ER positive (≥1%);
4. Premenopausal patients with age ≤35 years (at least menstruate once for prior 3 months, assess menstruation situation before chemotherapy if have);
5. No distant metastasis;
6. Clinical stage (TNM) meets at least one of the conditions as follow: T≥2cm or at least one region of regional lymph node metastasis (including micrometastases);
7. Patients must have undergone a surgery and (neo)adjuvant chemotherapy, targeted therapy, radiotherapy (if necessary) according to Chinese Anti-Cancer Association guidelines and specifications version 2015 for diagnosis and treatment of breast cancer;
8. Indexes of hematology and biochemistry conform to following standards: HGB≥10g/dl, WBC≥4,000/mm3, PLT≥100,000/mm3, GOT, GPT, ALP≤2xULN, TBIL, DBIL, CCr≤1.5xULN.

Exclusion Criteria:

1. Pregnant or lactating women or women of childbearing potential reject contraceptive measures;
2. History of organ transplantation (including autologous bone marrow transplantation and peripheral stem cell transplantation);
3. Concurrent malignancies or history of non-breast malignancies within the 5 years prior to study entry, except for curatively treated basal cell and squamous cell carcinomas of the skin, carcinoma in situ of the cervix; peripheral nervous system disorders caused by diseases or history of obvious mental and central nervous system disorders;
4. Prior use of neo-adjuvant chemotherapy after a definite diagnosis;
5. Nervous system disorders caused by diseases or obvious mental disorder, which would affect patients right to consent and compliance, or make patients in critical condition;
6. Serious hepatopathy (e.g., cirrhosis, etc.), nephropathy, respiratory illness, digestive illness or poorly controlled diabetes;
7. Cardiac illness with obvious abnormal EKG or clinical symptoms, namely congestive heart failure, coronary atherosclerotic heart disease with obvious symptoms, arrhythmia difficult to control by drugs, or history of myocardial infarction within the 12 months prior to study entry or class III/IV of cardiac function;
8. Concurrent treatment in another investigational trial;
9. Sensitivity or contraindication to any of the study medications.

Max Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 680 (Estimated)
Dates: Start 2016-03-30 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) | 5 years
  DFS is defined as the time between randomization and the date of the first occurrence of events as follow: local, regional recurrence or distant metastasis of invasive breast cancer, contralateral invasive breast cancer, or death due to any diseases. Patients who have not had disease progression or death at the end of follow-up (5 years) will be censored at the date last known to be alive and distant metastasis free. Subgroup analysis DFS of Luminal A and Luminal B breast cancer.

SECONDARY OUTCOMES:
Overall Survival (OS) | 5 years
  The time from randomization to death due to any cause. Patients still alive at the end of follow-up (5 years) will be censored at the last known alive date.
Invasive Breast Cancer Recurrence-Free Interval（BCFI) | 5 years
  The time between randomization and the first occurrence of local, regional recurrence or distant metastasis of invasive breast cancer, or contralateral invasive breast cancer. Patients who have not had invasive breast cancer recurrence at the end of follow-up (5 years) will be censored at the date last known to be distant metastasis free.
Adverse Effects Rate | 5 years

CONTACTS AND LOCATIONS:
Locations (24):
- China (24):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Peking University First Hospital, Beijing
  - Dongguan People's Hospital, Dongguan
  - GuangDong Hospital Of Traditional Chinese Medicine, Guangzhou
  - Guangdong People's Hospital, Guangzhou
  - Guangdong Provincial Women and Children's Hospital, Guangzhou
  - Guangzhou First Municipal People's Hospital, Guangzhou
  - Guangzhou Women and Childrens Medical Center, Guangzhou
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - Sun Yat-sen University Cancer Center, Guangzhou
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Guilin TCMhospital of China, Guilin
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Yunnan Cancer Hospital, Kunming
  - Maoming People's Hospital, Maoming
  - The first Affiliated Hospital of Guangxi Medical University, Nanning
  - The Affiliated Hospital of Qingdao University, Qingdao
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Affiliated hospital of Guangdong Medicine College, Zhanjiang
  - Lian Jiang People' s Hospital, Zhanjiang
  - Henan Cancer Hospital, Zhengzhou
  - Zhongshan People's Hospital, Zhongshan
  - The Fifth Affiliated Hospital Sun Yat-Sen University, Zhuhai

REFERENCES:
- [Background] Fan L, Strasser-Weippl K, Li JJ, St Louis J, Finkelstein DM, Yu KD, Chen WQ, Shao ZM, Goss PE. Breast cancer in China. Lancet Oncol. 2014 Jun;15(7):e279-89. doi: 10.1016/S1470-2045(13)70567-9. PMID 24872111
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Aromatase inhibitors versus tamoxifen in early breast cancer: patient-level meta-analysis of the randomised trials. Lancet. 2015 Oct 3;386(10001):1341-1352. doi: 10.1016/S0140-6736(15)61074-1. Epub 2015 Jul 23. PMID 26211827
- [Background] LHRH-agonists in Early Breast Cancer Overview group; Cuzick J, Ambroisine L, Davidson N, Jakesz R, Kaufmann M, Regan M, Sainsbury R. Use of luteinising-hormone-releasing hormone agonists as adjuvant treatment in premenopausal patients with hormone-receptor-positive breast cancer: a meta-analysis of individual patient data from randomised adjuvant trials. Lancet. 2007 May 19;369(9574):1711-23. doi: 10.1016/S0140-6736(07)60778-8. PMID 17512856
- [Background] Pagani O, Regan MM, Walley BA, Fleming GF, Colleoni M, Lang I, Gomez HL, Tondini C, Burstein HJ, Perez EA, Ciruelos E, Stearns V, Bonnefoi HR, Martino S, Geyer CE Jr, Pinotti G, Puglisi F, Crivellari D, Ruhstaller T, Winer EP, Rabaglio-Poretti M, Maibach R, Ruepp B, Giobbie-Hurder A, Price KN, Bernhard J, Luo W, Ribi K, Viale G, Coates AS, Gelber RD, Goldhirsch A, Francis PA; TEXT and SOFT Investigators; International Breast Cancer Study Group. Adjuvant exemestane with ovarian suppression in premenopausal breast cancer. N Engl J Med. 2014 Jul 10;371(2):107-18. doi: 10.1056/NEJMoa1404037. Epub 2014 Jun 1. PMID 24881463
- [Background] Francis PA, Regan MM, Fleming GF, Lang I, Ciruelos E, Bellet M, Bonnefoi HR, Climent MA, Da Prada GA, Burstein HJ, Martino S, Davidson NE, Geyer CE Jr, Walley BA, Coleman R, Kerbrat P, Buchholz S, Ingle JN, Winer EP, Rabaglio-Poretti M, Maibach R, Ruepp B, Giobbie-Hurder A, Price KN, Colleoni M, Viale G, Coates AS, Goldhirsch A, Gelber RD; SOFT Investigators; International Breast Cancer Study Group. Adjuvant ovarian suppression in premenopausal breast cancer. N Engl J Med. 2015 Jan 29;372(5):436-46. doi: 10.1056/NEJMoa1412379. Epub 2014 Dec 11. PMID 25495490